CLINICAL TRIAL: NCT03946293
Title: Increased Bioavailability of Phenolic Acids and Enhanced Vascular Function Following Intake of Feruloyl Esterase-processed High Fibre Bread: a Randomized, Controlled, Single Blind, Crossover Human Intervention Trial.
Brief Title: Enhanced Vascular Function Following Intake of Feruloyl Esterase-processed High Fibre Bread.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Biotechnology and Biological Sciences Research Council (Other)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor of Nutritional Medicine, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Wholegrain_FMD
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Cardiovascular Risk Factor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- White bread (Active Comparator): White bread 3 x 30 g, single serving
  Interventions: Dietary Supplement: White Bread
- Wholegrain (Active Comparator): Standard wholegrain, 3 x 30 g, single serving
  Interventions: Dietary Supplement: Wholegrain bread
- Wholegrain Enzyme (Experimental): Enzyme-treated wholegrain, 3 x 30 g, single serving
  Interventions: Dietary Supplement: Wholegrain Enzyme

INTERVENTIONS:
Dietary Supplement: White Bread — White bread made with commercial white flour with bran/fibre removed
  Arms: White bread
Dietary Supplement: Wholegrain bread — Wholegrain bread made with commercial wholegrain flour.
  Arms: Wholegrain
Dietary Supplement: Wholegrain Enzyme — Wholegrain bread made with enzyme-treated commercial wholegrain flour.
  Arms: Wholegrain Enzyme

SUMMARY:
This study evaluates the impact of a high phenolic acid intake from wholegrain wheat bread on human vascular function and plasma phenolic acid concentrations in healthy adults. All participants received a high fibre flatbread with enzymatically released free FA (14.22 mg), an equivalent standard high fibre bread (2.34 mg), or a white bread control (0.48 mg).

DETAILED DESCRIPTION:
Clinical trial data have indicated an association between wholegrain consumption and a reduction in surrogate markers of cardiovascular disease. A number of components of wheat have been suggested to contribute to the cardiovascular health benefits associated with wholegrain consumption, most notably the fiber component. However, phenolic compounds that are bound to arabinoxylan fibre, particularly the hydroxycinnamate ferulic acid, may also contribute, in part, to vascular health effects. These phenolics may be more active when released enzymatically from the fiber prior to ingestion.

The aim of the present study was therefore to determine whether the intake of high fibre bread containing higher free ferulic acid levels (enzymatically released during processing) enhances human endothelium-dependent vascular function to a greater extent than that of traditional wholegrain bread and/or a white bread control.

ELIGIBILITY:
Inclusion Criteria:

1) fasting lipids in the upper half of the normal range (triacylglycerol 0.8-3.2 mmol/l and total cholesterol 6.0-8.0 mmol/l); 2) BMI 25-32 kg/m2; 3) non-smoker; 4) not diabetic (diagnosed or fasting glucose < 7 mmol/l) or suffer from endocrine disorders; 5) hemoglobin and liver enzymes levels within the normal range [Alanine Transaminase (ALT): 0-55 IU/L; Alkaline Phosphatase (ALP): 38-126 U/L; Aspartate Transaminase (AST): 0-45 IU/L; Gamma Glutamyl Transferase (GGT): 12-58 IU/L]); 6) not having suffered a myocardial infarction/stroke in the past 12 months; 7) not suffering from renal or bowel disease or have a history of choleostatic liver or pancreatitis; 8) not on drug treatment for hyperlipidemia, hypertension, inflammation or hyper-coagulation; 9) not taking any fish oil, fatty acid or vitamin and mineral supplements; 10) no history of alcohol misuse; 11) not planning, or on a weight reduction regime; 12) not having taken antibiotics in the 6 months prior to the study; and 13) being able to consume the study interventions.

Exclusion Criteria:

* Gluten sensitive

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-11-15 (Actual)

PRIMARY OUTCOMES:
Flow-mediated dilatation (FMD) | Change from baseline to 5 hours
  FMD of the brachial artery

SECONDARY OUTCOMES:
Plasma phenolic acids | Change from baseline to 24 hours
  Presence of phenolic acid metabolites in the circulation over a 24 h period.
Laser Doppler Imaging with iontophoresis | Change from baseline to 5 hours
  Laser Doppler Imaging with iontophoresis (acetyl choline and sodium nitroprusside)
Digital Volume Pulse (DVP) | Change from baseline to 5 hours
  DVP stiffness index (DVP-SI) and DVP reflexion index (DVP-RI)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Food and Nutritional Sciences, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turner AL, Michaelson LV, Shewry PR, Lovegrove A, Spencer JPE. Increased bioavailability of phenolic acids and enhanced vascular function following intake of feruloyl esterase-processed high fibre bread: A randomized, controlled, single blind, crossover human intervention trial. Clin Nutr. 2021 Mar;40(3):788-795. doi: 10.1016/j.clnu.2020.07.026. Epub 2020 Aug 8. PMID 33077275